CLINICAL TRIAL: NCT00974818
Title: Mitomycin C Versus Bacillus Calmette-Guerin in the Intravesical Treatment of Non-Muscle-Invasive Bladder Cancer Patients: A Randomized Phase III Non-inferiority Trial
Brief Title: Mitomycin C Versus Bacillus Calmette-Guerin in the Intravesical Treatment of Non-Muscle-Invasive Bladder Cancer Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: New York Presbyterian Hospital (Other); Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-118
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Bladder Cancer
Keywords: Bladder; Mitomycin C; MMC; TheracysR Bacillus Calmette-Guerin; BCG; intravesical; 09-118
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Mitomycin; BCG Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pts getting Mitomycin C (MMC) (Experimental): Patients will receive a induction course of 6 cycles of weekly intravesical therapy of MMC, followed by a maintenance schedule consisting of 3 weekly cycles of the same drug at 3, 6, 12, 18, and 24 months.
  Interventions: Drug: Mitomycin C (MMC)
- pts getting Bacillus Calmette-Guerin (BCG) (Experimental): Patients will receive a induction course of 6 cycles of weekly intravesical therapy of either BCG, followed by a maintenance schedule consisting of 3 weekly cycles of the same drug at 3, 6, 12, 18, and 24 months.
  Interventions: Biological: Bacillus Calmette-Guerin (BCG)

INTERVENTIONS:
Drug: Mitomycin C (MMC) — Patients randomized to this group will receive six weekly cycles of 40 mg of intravesical MMC (dissolved in a total volume of 20 mL sterile water). Patients will receive three weekly cycles of 40 mg of intravesical MMC (dissolved in a total volume of 20 mL sterile water) 3, 6, 12, 18, and 24 months after the induction course.
  Arms: pts getting Mitomycin C (MMC)
Biological: Bacillus Calmette-Guerin (BCG) — Patients randomized to this group will receive six weekly cycles of 81 mg of intravesical BCG (dissolved in a total volume of 53 mL of diluent and saline). Patients will receive three weekly cycles of 27 mg of intravesical BCG (dissolved in a total volume of 53 mL of diluent and saline) 3, 6, 12, 18, and 24 months after the induction course.
  Arms: pts getting Bacillus Calmette-Guerin (BCG)

SUMMARY:
The purpose of this study is to compare the bladder cancer treatments, Mitomycin C (MMC) and Bacillus Calmette Guerin (BCG), to find out which is better. In this study, the patient will get either the Mitomycin C (MMC) or the Bacillus Calmette Guerin (BCG). They will not get both.

The patient had a Transurethral Resection (TUR) or an in office cystoscopy to make the diagnosis of bladder cancer. A biopsy was done and removed any tumors the doctor saw. Even after the doctor removes the tumors, the cancer can return. In this case, the doctor will put medicine into the bladder to destroy cancer cell. This is called intravesical therapy. The two most commonly used drugs for this purpose are MMC and BCG.

Both drugs have been studied for many years. They both show good results when compared to other treatments. They have not been studied using the schedule that will be used in the study. The doctor does not know if these two drugs are equally effective in treating the cancer and preventing recurrence.

BCG has been studied more often than MMC. The studies have shown that a long schedule of BCG is better than a short schedule of MMC. They have also shown that the side effects of BCG are more intense than with MMC. A recent study showed that a new dose of MMC is better than the old standard dose. Since the side effects of MMC occur less often, it is important to learn whether the two drugs are equally effective. That could help us decide between the treatments. In this study, the doctor will compare MMC and BCG when given for the same amount of time. The doctor hopes the study will tell us which drug is more effective in preventing the return of the cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Patients must have pathologically confirmed non-muscle invasive urothelial bladder carcinoma by the Department of Pathology New York Presbyterian Hospital, Weill Medical College of Cornell University or Memorial Sloan Kettering Cancer Center or a documented past history of Ta or T1 non-muscle invasive urothelial bladder tumors.
* Intermediate Risk UBC patients: Recurrence Total Score = 1 to 9

Exclusion Criteria:

* Any intravesical therapy within the past six months prior to current diagnosis
* Currently being treated or scheduled to have radiation treatment for bladder cancer during the study
* Scheduled to have surgery for bladder cancer during the study
* Currently being treated or scheduled to have treatment with any chemotherapeutic agent during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guido Dalbagni, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Weill Medical College of Cornell University, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Mitomycin C (MMC): Patients will receive a induction course of 6 cycles of weekly intravesical therapy of MMC, followed by a maintenance schedule consisting of 3 weekly cycles of the same drug at 3, 6, 12, 18, and 24 months.
  Mitomycin C (MMC): Patients randomized to this group will receive six weekly cycles of 40 mg of intravesical MMC (dissolved in a total volume of 20 mL sterile water). Patients will receive three weekly cycles of 40 mg of intravesical MMC (dissolved in a total volume of 20 mL sterile water) 3, 6, 12, 18, and 24 months after the induction course.
- Bacillus Calmette-Guerin (BCG): Patients will receive a induction course of 6 cycles of weekly intravesical therapy of either BCG, followed by a maintenance schedule consisting of 3 weekly cycles of the same drug at 3, 6, 12, 18, and 24 months.
  Bacillus Calmette-Guerin (BCG): Patients randomized to this group will receive six weekly cycles of 81 mg of intravesical BCG (dissolved in a total volume of 53 mL of diluent and saline). Patients will receive three weekly cycles of 27 mg of intravesical BCG (dissolved in a total volume of 53 mL of diluent and saline) 3, 6, 12, 18, and 24 months after the induction course.
Period: Overall Study
Arm/Group | Mitomycin C (MMC) | Bacillus Calmette-Guerin (BCG)
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mitomycin C (MMC) | Bacillus Calmette-Guerin (BCG) | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 8 | 19
  >=65 years | 14 | 17 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 20 | 21 | 41

OUTCOME MEASURES:

1. Primary Outcome: Response to Treatment
Description: will be assessed by cystoscopy every 3 months (+/- 3 weeks) in the first 2 years after induction.
Time Frame: 2 years
Population: Due to a lack of patients accrued to the protocol the protocol was closed and the analysis of the 2 year relapse rates could not be compared.
Measure: Number; unit: participants
Arm/Group | Mitomycin C (MMC) | Bacillus Calmette-Guerin (BCG)
Number analyzed (Participants) | 25 | 25
participants | 25 | 25

ADVERSE EVENTS:
Arm/Group | Mitomycin C (MMC) | Bacillus Calmette-Guerin (BCG)
Serious Adverse Events (participants affected / at risk) | 1/25 | 1/25
Other Adverse Events (participants affected / at risk) | 6/25 | 10/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mitomycin C (MMC) (N=25) | Bacillus Calmette-Guerin (BCG) (N=25)
Death not assoc w CTCAE term- Death NOS (General disorders) | 0 (0) | 1 (1)
Cystitis (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mitomycin C (MMC) (N=25) | Bacillus Calmette-Guerin (BCG) (N=25)
Cystitis (Renal and urinary disorders) | 4 (6) | 10 (12)
Pain - Penis (General disorders) | 2 (2) | 0 (0)
Urinary frequency/urgency (Renal and urinary disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes